CLINICAL TRIAL: NCT04728386
Title: Assessment of Postoperative Pain and Antibacterial Efficacy After Root Canal Irrigation With Curcumin Versus Sodium Hypochlorite in Patients With Necrotic Mandibular Molars: Randomized Clinical Trial
Brief Title: Postoperative Pain and Antibacterial Efficacy After Root Canal Irrigation With Curcumin or Sodium Hypochlorite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Medhat, post graduate student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CU-ENDO-11-10-2020
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Necrotic Pulp
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- curcumin irrigant (Experimental): final flush root canal irrigation with 5 ml curcumin solution
  Interventions: Other: curcumin solution
- sodium hypochlorite (Experimental): final flush root canal irrigation with 5 ml sodium hypochlorite
  Interventions: Other: sodium hypochlorite

INTERVENTIONS:
Other: curcumin solution — 2 % curcumin solution as root canal irrigant
  Arms: curcumin irrigant
Other: sodium hypochlorite — 2.5% sodium hypochlorite solution as root canal irrigant
  Arms: sodium hypochlorite

SUMMARY:
This study aims to compare the effect of 2% curcumin solution versus 2.5% sodium hypochlorite as irrigating solutions in necrotic mandibular molars in terms of postoperative pain and antibacterial effect.

DETAILED DESCRIPTION:
patients with necrotic mandibular molars will be selected

1. Diagnostic procedures:

   * Personal information (name, age, gender, address and phone number), full medical and dental histories using schematic charts will be obtained from all patients participating in this research.
   * History of chief complaint will be obtained in the dental history chart.
   * Clinical and radiographic evaluation for each tooth included in this study will be recorded. The tooth will be examined for presence of extensive caries or pulp exposures. Soft tissue examination and tooth mobility evaluation will be done by percussion and palpation.
   * Extraoral examination will be performed by visual inspection of the face and neck and palpation for any swollen lymph nodes.
   * Each tooth will be evaluated for sensitivity using electric pulp tester. Diagnosis will also be confirmed by the absence of bleeding after access cavity preparation.
   * Final Diagnosis: Mature mandibular asymptomatic necrotic molars with normal periapical radiographic appearance.
   * The operator will explicitly explain the trial steps to the patients, and an informed consent will be signed by patients who accept enrollment.
   * Pain scale chart will be given to each patient to rate his /her pain level before endodontic treatment as preoperative reading using a Numerical Rating Scale (NRS).
2. Endodontic procedures:

   * All the performed steps of root canal treatment will be included in the chart of endodontic procedures.
   * The tooth will be isolated with rubber dam to maintain aseptic field, after isolation the tooth and surrounding field will be disinfected by a protocol using 3% hydrogen peroxide and 2.5% sodium hypochlorite before and after coronal access cavity preparation.
   * The initial sample S1 will be collected from root canals before preparation using sterile paper points. Each root canal will be dried with 3 sterile paper points ISO# 15 which will be left inside the root canal for 1 minute each with pumping movements to generate a suspension with bacteria of the main pulpal area.
   * The paper points will be immediately placed in sterile test tubes containing reduced transport medium of thioglycolate and sent to the Microbiology Laboratory, Faculty of Medicine, Cairo University for microbiologic processing to be cultured within one hour.
   * Root canals will be mechanically prepared in a crown-down approach using ProTaper Universal NiTi files in an X-Smart endodontic motor according to the manufacture instructions.
   * The canals will be thoroughly irrigated between every two subsequent files using 2 ml of 2.5% NaOCl using a side vented needle (gauge 29) to control the possibility of irrigant apical extrusion.
   * After complete root canal preparation all canals will be flushed with 17 % EDTA followed by sterile saline.
3. Random allocation:

   * According to the randomization sequence, after complete root canal preparation patients will be assigned to one of 2 groups:

     * Intervention Group (G1): each canal will be flushed using 5 ml of curcumin solution in a plastic syringe with a side vented needle (gauge 29) inserted 1 ml shorter than the working length.
     * Comparator Group (G2): each canal will be flushed using 5 ml of 2.5% sodium hypochlorite in a plastic syringe with side vented needle (gauge 29) inserted 1 ml shorter than the working length.
   * After flushing the canals with each irrigating solution all canals will be flushed with 10 ml sterile saline and the final sample S2 will be collected in the same manner as S1 using sterile paper points ISO # 30/0.02 or # 40/0.02, corresponding to the size of the master apical file F3 or F4, respectively.
   * Root canals will be dried using ProTaper paper points. The root canals will be obturated using the modified single cone technique with resin based root canal sealer and ProTaper gutta-percha cones size F3 or F4 according to the size of the final finishing file, together with auxiliary cones ISO # 25/0.02.
   * After obturation, a cotton pellet will be placed in the pulp chamber and the access cavity will be sealed with a temporary filling.
   * All patients will be asked to record their postoperative pain level on Numerical Rating Scale (NRS) at 8, 24 and 48 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age between 18-50 years.
2. Male and female.
3. Systemically healthy patients (ASA I or II).
4. Mature mandibular molar teeth with: Necrotic pulps, normal periapical radiographic appearance and no intra-canal calcifications or internal resorptive lesions

Exclusion Criteria:

1. Medically compromised patients having substantive functional limitations (ASA III or IV).
2. Patients having two or more adjacent teeth requiring endodontic treatment.
3. Patients who received antibiotic therapy within the last three months before treatment.
4. Patients administered analgesics in the last 24 hours before treatment.
5. Teeth with:

   * Vital pulps.
   * Immature apices.
   * Acute periapical abscess, swellings and facial cellulitis.
   * Periodontally hopeless (mobility grade II or III).
   * Previous root canal treatment.
   * Non-restorable coronal portion.
6. TMJ problems, bruxism or traumatic occlusion.
7. Inability to perceive the given instructions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
postoperative pain at 8 hours | 8 hours
  recorded by 11-point NRS scale with scores from 0 to 10, with 0 for having no symptoms and 10 having worst imaginable symptoms. Pain levels will be categorized as follows:
  * 0 = no pain.
  * 1-3= mild pain.
  * 4-6= moderate pain.
  * 7-10= severe pain. scale with scores from 0 to 10, with 0 for having no symptoms and 10 having worst imaginable symptoms. Pain levels will be categorized as follows:
  * 0 = no pain.
  * 1-3= mild pain.
  * 4-6= moderate pain.
  * 7-10=severe pain
postoperative pain at 24 hours | 24 hours
  recorded by 11-point NRS scale with scores from 0 to 10, with 0 for having no symptoms and 10 having worst imaginable symptoms. Pain levels will be categorized as follows:
postoperative pain at 48 hours | 48 hours
  recorded by 11-point NRS scale with scores from 0 to 10, with 0 for having no symptoms and 10 having worst imaginable symptoms. Pain levels will be categorized as follows:

SECONDARY OUTCOMES:
antibacterial effect | during treatment
  assessment through culture and the count of Colony-Forming Units(CFUs)

CONTACTS AND LOCATIONS:
Overall Officials: eman medhat, Principal Investigator — Cairo University

REFERENCES:
- [Background] Yilmaz K, Tufenkci P, Adiguzel M. The effects of QMix and EndoActivator on postoperative pain in mandibular molars with nonvital pulps: a randomized clinical trial. Clin Oral Investig. 2019 Nov;23(11):4173-4180. doi: 10.1007/s00784-019-02856-6. Epub 2019 Feb 27. PMID 30815731
- [Background] Sotomil JM, Munchow EA, Pankajakshan D, Spolnik KJ, Ferreira JA, Gregory RL, Bottino MC. Curcumin-A Natural Medicament for Root Canal Disinfection: Effects of Irrigation, Drug Release, and Photoactivation. J Endod. 2019 Nov;45(11):1371-1377. doi: 10.1016/j.joen.2019.08.004. Epub 2019 Sep 18. PMID 31542283
- [Background] Purohit RN, Bhatt M, Purohit K, Acharya J, Kumar R, Garg R. Clinical and Radiological Evaluation of Turmeric Powder as a Pulpotomy Medicament in Primary Teeth: An in vivo Study. Int J Clin Pediatr Dent. 2017 Jan-Mar;10(1):37-40. doi: 10.5005/jp-journals-10005-1404. Epub 2017 Feb 27. PMID 28377653